CLINICAL TRIAL: NCT01582646
Title: Analgesic Effect of Beta 2-mimetics in the Treatment of Neuropathic Pain
Acronym: Bêtapain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulty of recruitment
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4705
Record Dates: First submitted 2012-04-10; First posted 2012-04-20 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Postthoracotomy Pain; Postthoracoscopy Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- first period with terbutaline and second period with placebo (Other): The studies will be randomized, double-blind, placebo-controlled. It will use a 4 + 4 weeks crossover design for terbutaline vs. placebo (no titration). A washout period (2 weeks) will separate the treatment periods.
  Interventions: Drug: Terbutaline sustained release 5 mg
- first period with placebo and second period with terbutaline. (Other): The studies will be randomized, double-blind, placebo-controlled. It will use a 4 + 4 weeks crossover design for terbutaline vs. placebo (no titration). A washout period (2 weeks) will separate the treatment periods.
  Interventions: Drug: Terbutaline sustained release 5 mg

INTERVENTIONS:
Drug: Terbutaline sustained release 5 mg — Terbutaline 10mg oral per day (5 mg twice a day) during 28 days

SUMMARY:
Neuropathic pain is due to a lesion or disease affecting the nervous system. Antidepressants (ADs) are recommended as the first line treatment. In a murine model, the investigators evidenced that antidepressants antiallodynic action is mediated through β2-adrenergic receptor stimulation and that β-mimetics display the same effect. These data support the idea that β-mimetics could offer a therapeutic alternative to ADs for neuropathic pain treatment. This study will aim at assessing the effects of terbutaline on neuropathic pain symptoms.

ELIGIBILITY:
Inclusion Criteria:

* adults from 18 to 75 years old
* neuropathic painful condition following a thoracotomy or thoracoscopy for at least 3 months

Exclusion criteria:

* cardiovascular risk
* unstable diabetes mellitus
* allergy for terbutaline
* hypokaliemia without treatment
* untreated hypothyroidism
* HIV- or chemotherapy-induced neuropathy
* cancer being treated by chemo- or radio-therapy
* concomitant treatment with β-blockers, tricyclic ADs or morphine
* concomitant pain more severe than neuropathic pain- pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average intensity of pain during the last 24 hours reported by the patient on a 11 points Numeric Scale | Day one, day 14 and day 28 of each 4 weeks period

CONTACTS AND LOCATIONS:
Overall Officials: André Muller, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (2):
- France (2):
  - CHU de Besançon, Besançon
  - Hôpitaux Universitaires de Strasbourg, Strasbourg